## Overcoming Barriers and Obstacles to Adopting Diabetes Devices

04161131

November 11, 2020

Molly Tanenbaum, Principal Investigator Stanford University Stanford, California 94305

## STATISTICAL ANALYSIS PLAN

For this pilot study we aimed to recruit between 20 and 40 adults with type 1 diabetes. Descriptive statistics were used to calculate frequencies and means for demographic and medical information. To examine changes from baseline to post-intervention in primary and secondary outcome variables, we used paired t-tests for normally distributed variables and Wilcoxon signed-rank tests for non-normally distributed variables. We then calculated effect sizes (Cohen's d; r). To assess feasibility and acceptability, we calculated percentage of eligible individuals who agreed to participate in the study, and percentage of participants who withdrew or were lost to follow-up. Focus group data was analyzed using content analysis.